CLINICAL TRIAL: NCT05282056
Title: COVID-19 Volumetric Quantification on Computer Tomography Using Computer Aided Diagnostics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogdan Bercean (Industry)
Collaborators: Pius Brinzeu Timisoara County Emergency Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Bogdan Bercean, Head of Artificial Intelligence, XVision
Organization: XVision (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 282/01.02.2022
Record Dates: First submitted 2022-03-14; First posted 2022-03-16 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: CAD; AI; Artificial Intelligence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: CAD outputs are turned off for randomly chosen 50% of patients, which represent the control group. The other 50% are analysed using CAD
Who Masked: Participant
Masking Description: The random assignment is done automatically by the CAD system and is not visible to the patient. The radiologist obviously sees which cases have CAD analysis and which not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD analysis (Experimental): The XVision COVID-19 computer aided diagnostic software is used by radiologist at CT analysis time
  Interventions: Diagnostic Test: CAD analysis
- No CAD analysis (No Intervention): No CAD analysis is shown to radiologist.

INTERVENTIONS:
Diagnostic Test: CAD analysis — CAD shows the radiologist automatically delineated areas of potential COVID-19 affection, together with an overall lung affection percentage.
  Arms: CAD analysis

SUMMARY:
The aim of the study is to asses the influence of computer aided diagnostic to the process of lung affection quantification on computer tomography in COVID-19 confirmed patients.

DETAILED DESCRIPTION:
The lung involvement of COVID-19 patients has been showed to be correlated to clinical outcomes and became part of the clinical practice. Even though various scores can be used, the affection estimation is usually done on computer tomography, using radiologists's estimation skills which is a highly subjective process.

Artificial intelligence is a known objective constant and therefore a potential radiologist complement. This trial aims at studying the effect of using a computer aided diagnostic software integrated in the normal clinical practice of radiologists from Timisoara County Emergency Hospital. It uses the AI-PROBE analysis setup, which turns off the CAD outputs for randomly chosen 50% the cases (control) and then compares the radiological reports for differences between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* RT-PCR confirmed patients of COVID-19

Exclusion Criteria:

* 15 or lower

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Mean difference of lung affection quantification percentage | At CT acquisition time, up to 2 weeks
  The objective measurement of lung affection percentage is measured against pixel level labels. A lower difference mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Pius Brinzeu Timisoara County Emergency Hospital, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Undecided
The statistical analysis, data points and possibly deidentified images.

REFERENCES:
- [Derived] Bercean BA, Birhala A, Ardelean PG, Barbulescu I, Benta MM, Rasadean CD, Costachescu D, Avramescu C, Tenescu A, Iarca S, Buburuzan AS, Marcu M, Birsasteanu F. Evidence of a cognitive bias in the quantification of COVID-19 with CT: an artificial intelligence randomised clinical trial. Sci Rep. 2023 Mar 25;13(1):4887. doi: 10.1038/s41598-023-31910-3. PMID 36966179